CLINICAL TRIAL: NCT01322048
Title: DASH After TBI Study: Decreasing Adrenergic or Sympathetic Hyperactivity After Severe Traumatic Brain Injury, A Pilot Randomized Clinical Trial Using Propranolol and Clonidine
Brief Title: DASH After TBI Study: Decreasing Adrenergic or Sympathetic Hyperactivity After Traumatic Brain Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Vanderbilt University Medical Center (Other); Eastern Association for the Surgery of Trauma (EAST) (Unknown)
Responsible Party: Principal Investigator, Mayur Patel, Assistant Professor of Surgery and Neurosurgery, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 110429
Record Dates: First submitted 2011-03-02; First posted 2011-03-24 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-07

CONDITIONS: Brain Injuries; Craniocerebral Trauma; Trauma, Nervous System; Traumatic Brain Injury
Keywords: Sympathetic Hyperactivity; Traumatic Brain Injury; Agitation; Severe TBI; TBI; Catecholamines; Heart rate variability; Adrenergic alpha-Agonists; Adrenergic beta-Antagonists; Cognitive Impairment
MeSH Terms: conditions — Brain Injuries; Craniocerebral Trauma; Trauma, Nervous System; Brain Injuries, Traumatic; Psychomotor Agitation; Cognitive Dysfunction | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adrenergic Blockade (Experimental): Propranolol and Clonidine
  Interventions: Drug: IV Propranolol and Per Tube Clonidine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IV Propranolol and Per Tube Clonidine — 1 mg IV q6h Propranolol and 0.1 mg Per Tube Clonidine, both for 7 days
  Arms: Adrenergic Blockade
Drug: Placebo — Placebo IV q6h and Per Tube q12, both for 7 days
  Arms: Placebo

SUMMARY:
The investigators intend to determine the effect of adrenergic blockade on 1) short-term physiology, behavior, and cognition and 2) long-term neuropsychological outcomes after severe Traumatic Brain Injury (TBI).

The primary hypothesis is that adrenergic blockade after severe TBI will be associated with increased ventilator-free days.

DETAILED DESCRIPTION:
Severe traumatic brain injury (TBI) is associated with sympathetic hyperactivity resulting in catecholamine excess, abnormal heart rate variability, agitation and sympathetic storms, deep white matter changes, and poor neuropsychological outcomes. Notably, persistent sympathetic hyperactivity after TBI results in higher days of mechanical ventilation and longer intensive care unit (ICU) length of stay (LOS). While there are data describing limited portions of this response, the full spectrum of sympathetic hyperactivity after severe TBI has not been systemically described or methodically intervened upon.

We will perform a double-blinded, randomized, placebo-controlled pilot trial in a 100 patient cohort in which one group will receive centrally acting sympatholytic drugs, propranolol and clonidine, and the other group, placebo, within 48 hours of severe TBI. The length of therapy will be 7 days.

The primary question studied is whether ventilator-free days will be increased after therapy.

Secondary endpoints include plasma and urine catecholamine levels, heart rate and blood pressure variability, responses to autonomic cold pressor testing, assessments of coma, sedation, and agitation, sedative requirements, analgesic use, antipsychotic medication use, coma-free days, ventilator-free days, Intensive Care Unit (ICU) length of stay, and survival. Also, neuropsychological outcomes will be measured at ICU discharge, 3 months, and 12 months.

Interim Analysis: At approximately 50% targeted accrual, n=46 randomized subjects, an interim analysis will be performed with A Priori (planned) futility and efficacy rules, which are DSMB and IRB approved.

ELIGIBILITY:
Inclusion Criteria:

* Age: 16 years to 64 years
* Glasgow Coma Scale score less than or equal to 8 (Severe TBI) with injury on CT
* Screen within 24 hours of injury

Exclusion Criteria:

* Pre-existing heart disease (i.e. coronary heart disease)
* Pre-existing cardiac dysrhythmia
* Allergy to study drugs
* Penetrating brain injury
* Pre-existing brain dysfunction (i.e. prior severe TBI, debilitating stroke)
* Impending brain herniation (i.e. loss of bilateral corneal reflexes)
* Craniectomy or craniotomy
* Spinal cord injury
* Myocardial injury
* Severe liver disease
* Current use of beta-blockers and/or alpha-2-agonist
* Withdrawal of care expected in 24 hours
* Prisoners
* Pregnant women
* Unable to follow-up through final visit

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2011-08; Primary Completion 2015-01 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mayur B Patel, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Nordness MF, Maiga AW, Wilson LD, Koyama T, Rivera EL, Rakhit S, de Riesthal M, Motuzas CL, Cook MR, Gupta DK, Jackson JC, Williams Roberson S, Meurer WJ, Lewis RJ, Manley GT, Pandharipande PP, Patel MB. Effect of propranolol and clonidine after severe traumatic brain injury: a pilot randomized clinical trial. Crit Care. 2023 Jun 9;27(1):228. doi: 10.1186/s13054-023-04479-6. PMID 37296432
- [Derived] Patel MB, McKenna JW, Alvarez JM, Sugiura A, Jenkins JM, Guillamondegui OD, Pandharipande PP. Decreasing adrenergic or sympathetic hyperactivity after severe traumatic brain injury using propranolol and clonidine (DASH After TBI Study): study protocol for a randomized controlled trial. Trials. 2012 Sep 26;13:177. doi: 10.1186/1745-6215-13-177. PMID 23013802
- See also: Vanderbilt Multidisciplinary Traumatic Brain Injury Clinic (MTBIC) — http://www.vanderbilthealth.com/traumasurvivors/36172

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject was enrolled but was not randomized/assigned to either arm, due to a late withdrawal of care decision.
Period: Overall Study
Arm/Group | Adrenergic Blockade | Placebo
Started | 21 | 26
Completed | 21 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adrenergic Blockade | Placebo | Total
Number analyzed (Participants) | 21 | 26 | 47
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 24 [21 to 34] | 27.5 [18.5 to 36] | 25 [19 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 16 | 25 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 26 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 19 | 24 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 26 | 47

OUTCOME MEASURES:

1. Primary Outcome: Ventilator-free Days
Time Frame: Baseline to day 28
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Adrenergic Blockade | Placebo
Number analyzed (Participants) | 21 | 26
days | 16.2 [5.5 to 20.1] | 18.05 [0.075 to 20.45]

2. Secondary Outcome: Plasma Norepinephrine Levels
Time Frame: Post-treatment (t=Day 8)
Population: Of those surviving treatment period
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Adrenergic Blockade | Placebo
Number analyzed (Participants) | 21 | 25
pg/mL | 962 [508 to 1471] | 714 [391 to 1257]

ADVERSE EVENTS:
Arm/Group | Adrenergic Blockade | Placebo
All-Cause Mortality (participants affected / at risk) | 5/21 | 8/26
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/26
Other Adverse Events (participants affected / at risk) | 0/21 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No